CLINICAL TRIAL: NCT00852137
Title: A Randomized, Double-blind, Vehicle-controlled Study to Evaluate the Pharmacokinetics of PEP005 (Ingenol Mebutate) Gel, 0.05%, When Applied in a Maximal Use Setting to the Dorsal Aspect of the Forearm in Patients With Actinic Keratosis
Brief Title: A Study to Evaluate the Pharmacokinetics of PEP005 (Ingenol Mebutate) Gel, 0.05%, When Applied in a Maximal Use Setting to the Dorsal Aspect of the Forearm in Patients With Actinic Keratosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peplin (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PEP005-017
Record Dates: First submitted 2009-02-22; First posted 2009-02-26 (Estimated); Results first posted 2012-05-28 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2012-04

CONDITIONS: Actinic Keratosis
Keywords: Peplin; PEP005; Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — 3-ingenyl angelate; Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEP005 (ingenol mebutate) Gel, 0.05% (Experimental)
  Interventions: Drug: PEP005 (ingenol mebutate) Gel, 0.05%
- Vehicle Gel (Placebo Comparator)
  Interventions: Drug: Vehicle Gel

INTERVENTIONS:
Drug: PEP005 (ingenol mebutate) Gel, 0.05% — PEP005 (ingenol mebutate) Gel 0.05% once daily for 2 consecutive days
  Arms: PEP005 (ingenol mebutate) Gel, 0.05%
Drug: Vehicle Gel — Vehicle Gel once daily for 2 consecutive days
  Arms: Vehicle Gel

SUMMARY:
This Phase II study is designed to evaluate the pharmacokinetics of PEP005 (ingenol mebutate) Gel, 0.05% when applied in a maximal use setting to the dorsal aspect of the forearm in patients with actinic keratoses

ELIGIBILITY:
Inclusion Criteria:

* Male or female;
* Multiple actinic keratosis (AK) lesions over a 100 cm^2 area of skin located on the dorsal aspect of one forearm.

Exclusion Criteria:

* Cosmetic or therapeutic procedures: within 2 weeks and within 2 cm of the selected treatment area(s);
* Treatment with immunomodulators, or interferon/interferon inducers or systemic medications that suppress the immune system: within 4 weeks;
* Treatment with 5-FU, imiquimod, diclofenac, or photodynamic therapy: within 8 weeks and within 2 cm of the selected treatment area(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Jarratt, MD, Principal Investigator — Derm Research, PLLC
Locations (1):
- DermResearch, Inc., Austin, Texas, United States

REFERENCES:
- [Derived] Anderson L, Jarratt M, Schmieder G, Shumack S, Katsamas J, Welburn P. Tolerability and Pharmacokinetics of Ingenol Mebutate 0.05% Gel Applied to Treatment Areas up to 100cm(2) on the Forearm(s) of Patients with Actinic Keratosis. J Clin Aesthet Dermatol. 2014 Dec;7(12):19-29. PMID 25584134
- See also: Food and Drug Authority — http://www.fda.gov

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Period:
  First patient randomized: March 18, 2009 Last patient completed Day 57: May 27, 2009 A single site in the US
Groups:
- PEP005 Gel, 0.05%: PEP005 (ingenol mebutate) Gel 0.05% once daily for 2 consecutive days
- Vehicle: Vehicle gel once daily for 2 consecutive days
Period: Overall Study
Arm/Group | PEP005 Gel, 0.05% | Vehicle
Started | 13 | 3
Completed | 13 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PEP005 Gel, 0.05% | Vehicle | Total
Number analyzed (Participants) | 13 | 3 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 2 | 10
  >=65 years | 5 | 1 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (9.7) | 64.7 (12) | 63.3 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 6 | 0 | 6
Region of Enrollment [Number; unit: participants]
  United States | 13 | 3 | 16

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Concentration (Cmax) for Ingenol Mebutate and Its Two Acyl Isomers (PEP015 and PEP025) Levels
Description: Maximum observed concentration (Cmax) for ingenol mebutate and its two acyl isomers (PEP015 and PEP025) levels over the 24 hour sampling time period based on actual values measured. Blood samples were taken: at 30 minutes, 1, 2, 4, 8, 12 and 24 hours following study medication application on Day 2.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PEP005 Gel, 0.05% | Vehicle
Number analyzed (Participants) | 13 | 3
ng/mL | NA (NA) — The assay results completed for the interim analysis, confirmed that there were no detectable levels of ingenol mebutate or its acyl isomers (PEP015 or PEP025) in any samples assayed. | NA (NA) — The assay results completed for the interim analysis, confirmed that there were no detectable levels of ingenol mebutate or its acyl isomers (PEP015 or PEP025) in any samples assayed.

2. Primary Outcome: Time at Which Cmax is Attained (Tmax) for Ingenol Mebutate, and Its Two Acyl Isomers (PEP015 and PEP025) Levels.
Description: Time at which Cmax is attained (Tmax) for ingenol mebutate, and its two acyl isomers (PEP015 and PEP025) levels measured at 30 min, 1, 2, 4, 8, 12 and 24 hours following study medication application on Day 2. If a maximum value occured at more than one timepoint Tmax is defined as the first timepoint with this value.
Time Frame: 1 day
Measure: Number; unit: hours
Arm/Group | PEP005 Gel, 0.05% | Vehicle
Number analyzed (Participants) | 13 | 3
hours | NA (NA) — The assay results completed for the interim analysis, confirmed that there were no detectable levels of ingenol mebutate or its acyl isomers (PEP015 or PEP025) in any samples assayed. | NA (NA) — The assay results completed for the interim analysis, confirmed that there were no detectable levels of ingenol mebutate or its acyl isomers (PEP015 or PEP025) in any samples assayed.

3. Primary Outcome: Area Under the Blood Conc. Versus Time Curve for Time 0-24 Hours (AUC(0-24)) for Ingenol Mebutate and Its Two Acyl Isomers (PEP015 and PEP025) Levels
Description: Area under the blood conc. versus time curve was calculated for time 0-24 hours (AUC(0-24)) for ingenol mebutate and its two acyl isomers (PEP015 and PEP025) levels measured at 30 min, 1, 2, 4, 8, 12 and 24 hours following study medication application on Day 2.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: ng/mL x h
Arm/Group | PEP005 Gel, 0.05% | Vehicle
Number analyzed (Participants) | 13 | 3
ng/mL x h | NA (NA) — The assay results completed for the interim analysis, confirmed that there were no detectable levels of ingenol mebutate or its acyl isomers (PEP015 or PEP025) in any samples assayed. | NA (NA) — The assay results completed for the interim analysis, confirmed that there were no detectable levels of ingenol mebutate or its acyl isomers (PEP015 or PEP025) in any samples assayed.

4. Secondary Outcome: Complete Clearance Rate in a 25 cm^2 Area Within the Selected Treatment Area
Description: Number of participants with complete clearence. Complete clearance rate is defined as no clinically visible actinic keratosis (AK) lesions in a 25 cm^2 area within the selected treatment area at Day 57 compared to baseline
Time Frame: baseline and day 57
Measure: Number; unit: participants
Arm/Group | PEP005 Gel, 0.05% | Vehicle
Number analyzed (Participants) | 13 | 3
participants | 10 | 0

5. Secondary Outcome: Percentage (%) Change in Actinic Keratosis (AK) Lesions in a 25 cm^2 Area Within the Selected Treatment Area
Description: Percentage (%) change in actinic keratosis (AK) lesions count at Day 57, compared to baseline, in a 25 cm^2 area within the selected treatment area.
Time Frame: Baseline and Day 57
Measure: Mean (Standard Deviation); unit: change from baseline lesion count (%)
Arm/Group | PEP005 Gel, 0.05% | Vehicle
Number analyzed (Participants) | 13 | 3
change from baseline lesion count (%) | -96 (8) | 33 (58)

6. Secondary Outcome: Number of Patients With Local Skin Responses (LSRs) Above 0 at Any Time Point During the Study.
Description: Number of patients with LSR at any time point during the study above 0. The treatment area was assessed at baseline and at each subsequent study visit for the presence and grade of the following Local Skin Responses (LSRs): erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, and erosion/ulceration using the Local Skin Response Grading Scale (version 5). Each LSR was graded from 0 (best outcome) to 4 (worst outcome). A composite LSR score was calculated as the sum of each individual LSR grade, giving a possible range of 0-24.
Time Frame: baseline and Day 2, 3, 8, 15, 29 and 57
Measure: Number; unit: participants
Arm/Group | PEP005 Gel, 0.05% | Vehicle
Number analyzed (Participants) | 13 | 3
participants | 13 | 1

7. Secondary Outcome: Patients With Incidence of Pigmentation and Scarring
Description: Patients with Incidence of pigmentation and scarring, and grade of pigmentation and scarring, following study treatment through Day 57
Time Frame: Baseline, Day 2, 3, 8, 15, 29 and 57
Measure: Number; unit: participants
Arm/Group | PEP005 Gel, 0.05% | Vehicle
Number analyzed (Participants) | 13 | 3
participants | 0 | 0

8. Secondary Outcome: Max Composite Local Skin Response (LSR) Score
Description: Max composite Local Skin Response (LSR) score on day 3 only . The treatment area was assessed at baseline and at each subsequent study visit for the presence and grade of the following Local Skin Responses (LSRs): erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, and erosion/ulceration using the Local Skin Response Grading Scale (version 5). Each LSR was graded from 0 (best outcome) to 4 (worst outcome). A composite LSR score was calculated as the sum of each individual LSR grade, giving a possible range of 0-24. (One vehicle treated patent had a LSR on day 1 only).
Time Frame: Day 3
Measure: Mean (Standard Deviation); unit: local skin response score
Arm/Group | PEP005 Gel, 0.05% | Vehicle
Number analyzed (Participants) | 13 | 3
local skin response score | 6.6 (3.1) | 0 (0)

ADVERSE EVENTS:
Time Frame: 57 days
Arm/Group | PEP005 Gel, 0.05% | Vehicle
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/3
Other Adverse Events (participants affected / at risk) | 3/13 | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PEP005 Gel, 0.05% (N=13) | Vehicle (N=3)
Toothache (Gastrointestinal disorders) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Evaluator and Principal Investigator agree not to individually publish the result of the study, but rather, to participate in a joint publication of the Study results coordinated by sponsor, who shall have the first righ to publish. If such joint publication is not submitted for publication within 1 year of study completion at all sites Evaluator and Principal Investigator have the right to individually produce and submit a proposed publication, subject to the prior review of sponsor.